CLINICAL TRIAL: NCT01313923
Title: Evaluation of Sirolimus for the Treatment of the Autoimmune Blistering Dermatosis Pemphigus
Brief Title: Evaluating Sirolimus to Treat Autoimmune Blistering Dermatosis Pemphigus
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Sergei Grando, MD, PhD, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-7844
Record Dates: First submitted 2011-03-10; First posted 2011-03-14 (Estimated); Results first posted 2016-03-25 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-05

CONDITIONS: Pemphigus
Keywords: Pemphigus
MeSH Terms: conditions — Pemphigus | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sirolimus (formerly known as Rapamycin) (Experimental): Subjects with stable pemphigus vulgaris already on treatment with prednisone will be enrolled. Subjects will start taking oral sirolimus and have it up-titrated while decreasing the prednisone dosage. Their disease state will be monitored during this time.
  Interventions: Drug: Sirolimus (formerly known as Rapamycin)

INTERVENTIONS:
Drug: Sirolimus (formerly known as Rapamycin) — For low to moderate immunologic risk, the loading dose is 6mg immediately after transplantation, followed by 2mg PO Qday in conjunction with cyclosporine and corticosteroids. After 2-4 months, cyclosporine should be discontinued over 4-8 weeks while titrating sirolimus drug concentrations within the target-range with whole blood trough concentrations every 1-2 weeks. Monitoring is needed because cyclosporine inhibits the metabolism of sirolimus, and discontinuation of cyclosporine can lead to lower levels of sirolimus. In high immunologic risk patients, the loading dose is 15mg after transplantation, followed by 5mg PO Qday in conjunction with cyclosporine and corticosteroids for 12 months. A whole blood trough level is recommended between days 5 and 7 with adjustment to the daily dose.
  Other Names: Sirolimus; Rapamycin

SUMMARY:
The purpose of this research is to study alternative treatments for the skin disease pemphigus (a rare autoimmune blistering disorder of the skin) by using sirolimus, an immunosuppressive drug. Immunosuppressive drugs inhibit or prevent the activity of the immune system and are commonly used to treat autoimmune diseases, inflammatory diseases, and organ transplantation rejection.

DETAILED DESCRIPTION:
The purpose of this study is to explore a new medication for the skin disease termed pemphigus. Our specific aim is to determine whether the use of sirolimus will allow for a decrease in the dosage or possibly eliminate the need for corticosteroids, which so far is the only type of drug that can control this disease.

Pemphigus is an autoimmune disease characterized by blistering, caused by autoantibodies against certain cells in the skin. This disease most commonly occurs in individuals ages 50 and older, and it presents as painful shallow erosions and/or blisters in the mouth and/or skin. Pemphigus is very painful and uncomfortable, associated with impaired quality of life and significant morbidity. Severe or untreated cases of pemphigus can become fatal if the involved surface area becomes large enough to cause dehydration and/or infection. The first line of therapy, and the standard of care, for pemphigus remain to be systemic corticosteroids. However, corticosteroids have many known side effects, especially when used for a long time. Many cases of pemphigus are insufficiently controlled with corticosteroids alone and require the addition of other immunosuppressive agents, such as azathioprine, cyclophosphamide, mycophenolate mofetil, or a variety of other therapies used off-label. All of these treatments are not always successful and have undesirable side effects, including increased risk of malignancy and infections. Although these treatments can offer some relief from the disease, they are also often the cause of many side effects.

Sirolimus (formerly known as rapamycin) is a drug commonly used after renal transplants to prevent organ rejection. In this study, pemphigus subjects with active disease will begin taking sirolimus in conjunction with corticosteroids, using a similar regimen used for organ transplantation to treat pemphigus. While increasing sirolimus and decreasing the corticosteroids, subjects will be monitored over a 12 month period to evaluate their disease response. The purpose of this study is to observe data trends.

Our specific aim is to determine whether the use of sirolimus will allow for a decrease in the dosage of the corticosteroid prednisone, which so far is the only type of drugs that can control these diseases, without making the pemphigus worse.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be 18 years of age or older.
2. Subject must have an established diagnosis of pemphigus disorder via biopsy and/or serologic titer, as determined appropriate by the lead researcher.
3. Subject must have active disease at the time of enrollment, as defined by a positive Nikolsky sign.
4. Subject must not be taking any immunosuppressive medication or therapy other than corticosteroids.
5. Subject must be able to understand and follow directions.
6. If female, subject is not currently breast feeding and/or pregnant as confirmed via negative pregnancy test, no potential for pregnancy, or if of child-bearing age, agrees to using birth control for entire duration of study and 12 weeks after end of study.

Exclusion Criteria:

1. Subject may not be under 18 years old.
2. Subject cannot understand or follow directions.
3. Subject may not have any condition that could, in the opinion of the investigator, compromise the subject's ability to give written consent and/or comply with the study procedures, such as a history of substance abuse or a psychiatric condition.
4. If female and of child bearing age, is pregnant or unwilling to use birth control during the study period.
5. Subject may not have any of the following laboratory abnormalities at baseline:

   * total white blood cell count < 2,000/mm3 or platelet count < 100,000/mm3
   * creatinine >1.5mg/dL
   * urine analysis protein of 2+ or greater
   * fasting triglycerides > 400 mg/dL, fasting total cholesterol > 300 mg/dL, or fasting LDLcholesterol > 160 mg/dL
   * transaminases > 2 times the upper limit of normal
6. Subjects may not be using any of the following medications: systemic antifungals, antiepileptics, HIV protease inhibitors, cimetidine, cisapride, clarithromycin, danazol, diltiazem, erythromycin, metoclopramide, rifabutin, rifampin, rifapentine, troleandomycin, or verapamil
7. Subject may not consume grapefruit juice and/or St. John's Wort (hypericum perforatum) throughout the duration of the study.
8. Subject may not have other significant concurrent medical conditions, including

   * Active malignancy, including evidence of cutaneous basal or squamous cell carcinoma or melanoma, or history of cancer (other than fully resected and surgically cured cutaneous basal cell and squamous cell carcinoma) within 5 years before the first 13 of 25 sirolimus dose. If malignancy occurred more than 5 years ago, documentation of disease-free state since treatment is required.
   * Known immunodeficiency syndromes, including HIV
   * Renal failure or insufficiency, as defined by laboratory parameters above
   * Significant proteinuria, as defined by laboratory parameters above
   * History of high cholesterol, lipids, or liver disease, as defined by laboratory parameters above
   * Uncontrolled hypertension, as defined by a blood pressure > 140/90 despite optimal medical therapy, as prescribed by primary care doctor
   * Any condition that, in the opinion of the investigator, might cause this study to be detrimental to the subject
   * Any active Common Terminology Criteria (CTC) grade 2 (localized infection; requiring local intervention) or higher infection (including chronic or localized infections) within 30 days prior to screening, at screening, or during screening period prior to first dose of sirolimus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergei Grando, MD, PhD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: three patients were screened and enrolled in the study.
Pre-assignment Details: Only major consideration for the pre-assignment is to exclude any patient with underlying immunodeficiency or hematological disorder. Investigational product itself can suppress hematopoiesis and is an immuno-modulator.
  All three patients screened were enrolled in the study.
Groups:
- Sirolimus: There is one arm to the study. All patients will be open-label, Sirolimus. There is no set dosage: medication dose will be based on FDA approved guidelines.
Period: Overall Study
Arm/Group | Sirolimus
Started | 3
Completed | 0
Not Completed | 3
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Groups:
- Sirolimus: All patient will be open-label; Sirolimus. Dosage is variable based on FDA guidelines.
Arm/Group | Sirolimus
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 59 [57 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Improvement of ABSIS Score While Reducing Steroid Dosage
Description: Measurement of disease severity will be quantified using ABSIS (Autoimmune Bullous Skin Disorder Intensity Score). Improvement in disease control is quantified by the maintenance or improvement of ABSIS score while reducing steroid dosage.
  No results as study has been terminated early by the investigator.
Time Frame: Expected time line 24 months
Population: This outcome was not assessed because no participant completed any visits of the study
Groups:
- Sirolimus (Formerly Known as Rapamycin): No results. Study has been terminated by investigator.
Arm/Group | Sirolimus (Formerly Known as Rapamycin)
Number analyzed (Participants) | 0

2. Secondary Outcome: Statistical Measures
Description: The statistical goal is to observe "success," an improvement in disease control while up-titrating sirolimus dosage. As there will be no control group, the subject or progress at the end of the study will be compared to their baseline at the beginning of the study. The subject and disease severity at the beginning of the study will be compared to the disease severity at each visit and be correlated with the dosage of sirolimus and corticosteroid. However, since no patient completed the study, the outcome and any data collected was not assessed.
Time Frame: Study early termination by investigator - no participant completed any visits of the study - no measurements taken
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Serious and Other (Not Including Serious) Adverse Events were not collected/assessed
Groups:
- Sirolimus (Formerly Known as Rapamycin): No results as study has been terminated early by the investigator.
Arm/Group | Sirolimus (Formerly Known as Rapamycin)
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
No results as study has been terminated early by the investigator.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No